CLINICAL TRIAL: NCT06992466
Title: Short Term Outcomes After Primary PCI in Diabetic Patients Treated With Insulin Versus Oral Anti-diabetic Drugs
Acronym: Observ
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walid shehata ahmed, doctor, Assiut University
Other Study IDs: Diabetic patients after PPCI
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus; PCI
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oral diabetic drugs: insulin

SUMMARY:
• This study aims to compare the short-term clinical and echocardiographic outcomes of primary PCI in diabetic patients treated with insulin versus OADs.

DETAILED DESCRIPTION:
1. Diabetes mellitus (DM) is a major risk factor for cardiovascular disease (CVD), significantly increasing the risk of myocardial infarction (MI), heart failure, and mortality. Among patients with ST-segment elevation myocardial infarction (STEMI), diabetes is associated with higher rates of multi vessel disease, impaired coronary microcirculation, and poorer outcomes following percutaneous coronary intervention (PCI) compared to non-diabetic patients (1.2.3.4)
2. Diabetes is an independent risk factor for the development of CAD. Coronary arteries in diabetic patients present extensive and diffuse atherosclerosis, longer and more complex lesions than in non-diabetic patients [5]. The relative risk of myocardial infarction (MI) is 50% higher in diabetic men and 150% higher in diabetic women [6]. Patients with type 2 DM have similar risk for cardiac events as subjects with a prior MI [7]. The risk of recurrence of MI in diabetic patients is more than 40% [8]. Due to high prevalence of acute MI in diabetic patients, adults with diabetes will lose 30 quality-adjusted life years compared to those without DM [9].
3. Primary PCI is the gold-standard treatment for STEMI, offering superior outcomes compared to fibrinolysis. However, diabetic patients exhibit higher rates of in-stent restenosis, stent thrombosis, and recurrent ischemic events, making optimal glycemic control and choice of anti-diabetic therapy critical in improving post-PCI outcomes (10)
4. Cardiac remodeling refers to a spectrum of structural and functional changes that occur in the heart in response to myocardial injury or increased hemodynamic load, such as after myocardial infarction, chronic hypertension, or valvular heart disease. These changes may include alterations in ventricular size, shape, wall thickness, and overall function, and they are strongly associated with adverse cardiovascular outcomes including heart failure and sudden cardiac death.

   Echocardiography is a cornerstone non-invasive imaging modality that plays a vital role in the assessment and monitoring of cardiac remodeling. It offers real-time evaluation of cardiac chamber dimensions, wall thickness, ventricular volumes, ejection fraction, myocardial deformation (strain), and diastolic function. These echocardiographic parameters not only reflect the extent of remodeling but also have prognostic significance in various cardiac conditions.(11)
5. Impact of Diabetes Treatment on Cardiovascular Outcomes

The choice of anti-diabetic therapy may influence cardiovascular outcomes in STEMI patients undergoing PCI. There are two main therapeutic strategies for diabetes management:

Insulin therapy: Often used in patients with long-standing or poorly controlled diabetes, but is associated with increased risks of hypoglycemia, weight gain, and potential pro-inflammatory effects, which may contribute to worse cardiovascular outcomes (12.13)

Oral anti-diabetic drugs (OADs): Certain newer agents, such as SGLT2 inhibitors and GLP-1 receptor agonists, have demonstrated cardio protective effects, while others like sulfonylureas may be associated with an increased risk of adverse cardiovascular events (14)

Despite these differences, data on the impact of insulin versus OADs on PCI outcomes remain inconclusive, necessitating further research

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM (type 2) undergoing primary PCI for STEMI.1-

Treated with either insulin or OADs prior to admission.2-

3- Age ≥18 year

Exclusion Criteria:

* Type 1 DM.1- Patients on both insulin and OADs.2- 3-Prior coronary artery bypass graft (CABG) surgery. 4-Severe renal impairment (eGFR <30 mL/min/1.73m²). 5-Hemodynamically unstable patients 6-moderate to severe VHD 7-Patients who were shifted from OADs to insulin during Follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 210 patients fulfilling our criteria presenting to emergency room of Assiut University hospitals. Patients will be involved in the study after obtaining a written informed consent and after approval of the faculty of medicine ethics committee.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Short Term Outcomes after Primary PCI in Diabetic Patients Treated with Insulin Versus Oral Anti-diabetic Drugs | baseline
  To compare major adverse cardiovascular events (MACE) in insulin-treated versus OAD-treated diabetic patients undergoing primary PCI.

SECONDARY OUTCOMES:
Echocardiography | baseline
  Echocardiographic assessment of cardiac Remodeling early and 3 months post primary PCI

CONTACTS AND LOCATIONS:
Overall Officials: ahmed, Study Director — Assiut University
Locations (1):
- Assuit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Background] Abizaid A, Kornowski R, Mintz GS, Hong MK, Abizaid AS, Mehran R, Pichard AD, Kent KM, Satler LF, Wu H, Popma JJ, Leon MB. The influence of diabetes mellitus on acute and late clinical outcomes following coronary stent implantation. J Am Coll Cardiol. 1998 Sep;32(3):584-9. doi: 10.1016/s0735-1097(98)00286-1. PMID 9741497
- [Background] Haffner SM, Lehto S, Ronnemaa T, Pyorala K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in nondiabetic subjects with and without prior myocardial infarction. N Engl J Med. 1998 Jul 23;339(4):229-34. doi: 10.1056/NEJM199807233390404. PMID 9673301